CLINICAL TRIAL: NCT05324046
Title: Comparison of Low Dose Contrast Enhanced Abdominal CT With Deep Learning Reconstruction With Standard Dose CT With Iterative Reconstruction in Patients With Suspected Liver Metastases: A Prospective Multicenter Study
Brief Title: Comparison Between LDCT With DL Recontruction and Standard Dose CT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: 2022-0410
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Liver Metastases
Keywords: CT; metastasis; liver
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver metastasis: Patients with suspicion of liver metastasis and scheduled for CT
  Interventions: Diagnostic Test: contrast-enhanced abdomen CT

INTERVENTIONS:
Diagnostic Test: contrast-enhanced abdomen CT — contrast-enhanced abdomen CT using dual-source CT scanner using A-tube (67% radiation) and B-tube (33% radiation).
  * full dose CT data (A +B tubes, 100%) are reconstructed with iterative reconstruction (conventional)
  * low dose CT data (A-tube only, B-tube only) are reconstructed with deep learning commercially available software.
  * images are reconstructed using full dose (A- & B- tubes) and smaller dose (A-tube only, B-tube only)

SUMMARY:
This prospective study aims to perform intra-individual comparison of the image quality between low dose liver CT with deep learning reconstruction and standard dose liver CT with iterative reconstruction in patients with liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* patients with underlying malignancy and suspicion of liver metastasis
* patients with known liver metastasis and on follow-up
* AND scheduled for contrast enhanced abdomen CT
* signed informed consent

Exclusion Criteria:

* absolute or relative contra-indication for contrast-enhanced CT
* diffuse infiltrative liver lesion or multiple (> 10) metastases

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred to Radiology department for undergoing contrast-enhanced abdomen CT.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
liver lesion conspicuity | 6 months after the CT scan
  graded on a five-point scale (1-5) with higher score indicates a better conscpicuity.

SECONDARY OUTCOMES:
liver lesion detectability | 6 months after the CT scan
  liver lesion detection rate on standard dose CT and low dose CT by blinded reviewers

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee TY, Yoon JH, Park JY, Park SH, Kim H, Lee CM, Choi Y, Lee JM. Intraindividual Comparison of Image Quality Between Low-Dose and Ultra-Low-Dose Abdominal CT With Deep Learning Reconstruction and Standard-Dose Abdominal CT Using Dual-Split Scan. Invest Radiol. 2025 Jul 1;60(7):454-462. doi: 10.1097/RLI.0000000000001151. Epub 2025 Jan 28. PMID 39874436